CLINICAL TRIAL: NCT03945890
Title: Health Management Center, Far Eastern Memorial Hospital
Brief Title: Importing Quality Improvement Practices and Enhance Health Education to Improving Quality of Bowel Preparation
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chen-Shuan Chung, Gastroenterologist, Division of Gastroenterology and Hepatology, Far Eastern Memorial Hospital
Other Study IDs: 104107-E
Record Dates: First submitted 2019-04-18; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: No-Show Patients
Keywords: quality improvement; team resource management; bowel preparation; health screening colonoscopy
MeSH Terms: conditions — No-Show Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Importing quality improvement practices and enhances health education to improving quality of bowel preparation for health screening colonoscopy

This is a retrospective data analysis study aimed at obtaining the types of purgative treatments used, the results of bowel preparation, and each subject's demographic characteristics (Age & Gender).

DETAILED DESCRIPTION:
This study aimed to check-up the result and the impact of patient education using a medical team resource management (TRM) method on the adequacy of bowel preparation.

Investigators collected a total of 2,104 (884 female, 1,220 male) healthy subjects who underwent a health check-up colonoscopy screening were enrolled before and after the application of the TRM program intervention. The efficacy of the TRM intervention and the factors affecting bowel preparation were estimated using multivariate logistic regression in this study.

Enrollment of study subjects and data collection: The subjects enrolled in this study were those who received a health check-up colonoscopy screening in a tertiary center, Far Eastern Memorial Hospital (FEMH), in Taiwan from March 2013 to August 2014. A total of 2,104 healthy subjects who underwent check-up colonoscopy screening were enrolled during the pre-intervention, post-intervention, and validation periods. Investigators need to collect each subject's demographic characteristics (Age & Gender) and the types of purgative treatments used were collected to analyze. According to the Aronchick Bowel Preparation Scale, this study divided the degree of bowel cleansing into four levels, namely, "Excellent", "Good", "Fair" and "Poor". Investigators also need to collect the results of bowel preparation to calculate of the adequate bowel cleansing rate was defined further as the percentage of the participants with "Excellent" or "Good" cleansing in our analysis.

ELIGIBILITY:
Inclusion Criteria:

* The healthy population who received a health check-up colonoscopy screening in Far Eastern Memorial Hospital (FEMH)
* Exam date from March 2013 to August 2014
* Age from 20 y/o to 80 y/o

Exclusion Criteria:

* Gastroenterology outpatients/inpatients
* Missing data subjects
* Out of the Age limits subjects
* Out of the Time period subjects

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study was secondary data analysis, and the data contains no person's details, images, or videos.
Study Population: This study was secondary data analysis, and the data contains no person's details, images, or videos. This is a retrospective data analysis study, investigators collected data enrolled in this study were those who received a health check-up colonoscopy screening in a tertiary center hospital, Far Eastern Memorial Hospital (FEMH), in Taiwan from March 2013 to August 2014. A total of 2,104 healthy subjects who underwent check-up colonoscopy screening were enrolled during the pre-intervention, post-intervention, and validation periods. Each subject's demographic characteristics (Age & Gender) and the type of purgative treatments used were collected. And health screening Bowel Preparation Scale including "Excellent", "Good", "Fair" and "Poor".
Sampling Method: Non-Probability Sample
Enrollment: 2104 (Actual)
Dates: Start 2015-09-12 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
The well-designed education intervention can improve the rate of adequate bowel pr eparation for health screening colonoscopy. | From March 2013 to August 2014.
  The multivariate logistic regression analysis results for adequate bowel preparation after adjustments for age, gender, purgative type, to analyze the adequate bowel preparation rate with different intervention period.
  Bowel preparation rate were the Good & Excellent % of the total cases. Each subject's demographic characteristics (Age & Gender), the type of purgative and bowel preparation rate were collected from Far Eastern Memorial Hospital (FEMH) in Taiwan. This study was secondary data analysis, and the data contains no person's details, images, or videos. This is a retrospective data analysis study, investigators collected data enrolled in this study were those who received a health check-up colonoscopy screening.

CONTACTS AND LOCATIONS:
Locations (1):
- Oriental Institute of Technology / Far Eastern Memorial Hospital, New Taipei City, Pan-Chiao Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung CS, Lin CM, Chen MS. Quality Improvement of Bowel Preparation for Screening Colonoscopies: A Study of Hospital Team Resource Management in Taiwan. Qual Manag Health Care. 2021 Apr-Jun 01;30(2):127-134. doi: 10.1097/QMH.0000000000000310. PMID 33783425